CLINICAL TRIAL: NCT02158195
Title: Immunopathology of Autoimmune Hemolytic Anemia: an Open, Prospective and Multicenter Study
Brief Title: Immunopathology of Autoimmune Hemolytic Anemia
Acronym: IAHAI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: AUDIA APJ 2012
Record Dates: First submitted 2014-03-05; First posted 2014-06-06 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Autoimmune Hemolytic Anemia
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Patients
  Interventions: Biological: blood samples
- controls
  Interventions: Biological: blood samples

INTERVENTIONS:
Biological: blood samples

SUMMARY:
Autoimmune hemolytic anemia (AIHA) is an auto-immune disease mediated by specific antibodies targeting red blood cells. Its pathogenesis is not completely understood, and the role of T cells have been rarely studied.

The aim of this study is to compare the frequency of circulating T cells, T cell polarization and functions, notably regulatory T cells, during warm AIHA by comparison to healthy controls.

The role of treatments, such as steroids, will also be determined in patients with warm AIHA.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with primary warm Autoimmune Hemolytic Anemia (wAIHA)
* Secondary AHAI (infections, hematological diseases, systemic diseases)
* Naive of treatment for hemolytic anemia or in relapse
* Older than 16
* Able to understand written and spoken French
* who have provided written informed consent
* INCLUSION CRITERIA for CONTROLS
* Persons without auto-immune disease, cancer or active infection.
* Older than 16
* Able to understand written and spoken French
* who have provided written informed consent

Exclusion Criteria:

* Cold agglutinin disease
* Pregnancy
* Persons without national health insurance

Exclusion Criteria for Controls:

* Subjects treated with corticosteroids or immunosuppressants
* Pregnancy
* Persons without national health insurance

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with warm primary or secondary Autoimmune Hemolytic Anemia
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2013-07-03 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2018-12-27 (Actual)

PRIMARY OUTCOMES:
physiological parameter : blood level of regulatory T cells (Treg, CD4+CD25HighFoxp3+) | Change from baseline to 3 months
physiological parameter : percentage of inhibiting LT proliferation inhibition | Change from baseline to 3 months

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHU de Besançon, Besançon
  - CH de Chalon-sur-Saône, Chalon-sur-Saône
  - CHU de DIJON, Dijon
  - CH de Mâcon, Mâcon
  - CH de METZ, Metz

REFERENCES:
- [Result] Ciudad M, Ouandji S, Lamarthee B, Cladiere C, Ghesquiere T, Nivet M, Thebault M, Boidot R, Soudry-Faure A, Chevrier S, Richard C, Maillet T, Maurier F, Greigert H, Genet C, Ramon A, Trad M, Predan V, Saas P, Samson M, Bonnotte B, Audia S. Regulatory T-cell dysfunctions are associated with increase in tumor necrosis factor alpha in autoimmune hemolytic anemia and participate in Th17 polarization. Haematologica. 2024 Feb 1;109(2):444-457. doi: 10.3324/haematol.2023.282859. PMID 37534543
- [Derived] Audia S, Bach B, Samson M, Lakomy D, Bour JB, Burlet B, Guy J, Duvillard L, Branger M, Leguy-Seguin V, Berthier S, Michel M, Bonnotte B. Venous thromboembolic events during warm autoimmune hemolytic anemia. PLoS One. 2018 Nov 8;13(11):e0207218. doi: 10.1371/journal.pone.0207218. eCollection 2018. PMID 30408135